CLINICAL TRIAL: NCT07222891
Title: Validating the Impact of Smell Testing on Health Outcomes and Provider Engagement.
Brief Title: Impact of Smell Testing on Health Outcomes
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Monell Chemical Senses Center (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Valentina Parma, Assistant Member and Senior Director of Multisector Engagements, Monell Chemical Senses Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 856831; R44DC022498 (NIH)
Record Dates: First submitted 2025-10-22; First posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Olfactory Dysfunction; Wellbeing
Keywords: Olfactory testing; Smell dysfunction; Psychological health; Randomized clinical trial; Patient-centered care; Access to care
MeSH Terms: conditions — Olfaction Disorders; Psychological Well-Being | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Olfactory data will be collected with six standardized smell tests in the in-person cohort and four standardized smell tests in the remote cohort. The research team will assess odor detection, intensity, identification, pleasantness and discrimination. Based on the cut-off scores determined before the beginning of data collection, the investigators will assign a participant to the smell dysfunction group or to the normosmia (non-smell dysfunction) group. Based on this diagnostic intervention, participants with smell dysfunction will receive patient-centered information and education about i) community engagement with individuals with smell loss, ii) available counseling and iii) medical support.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smell dysfunction detection and educational intervention (Experimental): Participants will take smell tests and receive educational materials on smell dysfunction.
  Interventions: Behavioral: Patient-centered information and education
- Normosmia (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Patient-centered information and education — Participants with smell dysfunction will receive patient-centered information and education about i) community engagement with individuals with smell loss, ii) available counseling and iii) medical support.
  Arms: Smell dysfunction detection and educational intervention

SUMMARY:
Smell dysfunction is frequent yet neglected. The sense of smell plays a crucial role in signaling disease, safety, and overall quality of life. However, the significance of a functional sense of smell in terms of health and well-being is often overlooked until one experiences a loss of smell due to injury or disease. Research demonstrates that individuals are often not self-aware of their smell dysfunction (i.e. they do not spontaneously report smell dysfunction as a symptom), especially if the changes are gradual, as in normal aging. Patients with smell dysfunction experience a marked reduction in quality of life, poor mental health, nutritional health, and brain health as well as increased 5- and 10-year mortality in older adults. This study explores whether or not enabling healthcare providers to offer resources and guidance on coping strategies for smell dysfunction improves health and wellbeing in those who experience it.

DETAILED DESCRIPTION:
The investigators will recruit participants in cycles for in person or remote participation. Each cycle is characterized by an initial assessment, intervention deployment (smell testing), post-intervention evaluation, 1-month and 6-month follow-ups via survey, text or phone to assess post-intervention psychological health and connection to care for smell dysfunction. The research team will assess odor detection, intensity, identification, pleasantness and discrimination. Based on the cut-offs determined prior to the beginning of data collection, the investigators will prospectively assign a participant to the smell dysfunction group or to the normosmia (no smell dysfunction) group. Based on this diagnostic intervention, participants with smell dysfunction will receive patient-centered information and education about i) community engagement with individuals with smell loss, ii) available counseling and iii) medical support. At the end of the 1-month and 6-month follow-up periods, the investigators will assess effectiveness of the intervention using pre-post comparisons to determine whether individuals taking a smell test felt improvements in their psychological health and whether they have contacted a provider and/or followed up with a visit.

Sessions may include multiple surveys/instruments depending on the session number. Specifically, emotional ratings and demographic information will be collected by means of either a paper - or computer-based questionnaire. A survey to measure psychological health and quality of life will be given to participants, as well as a questionnaire to measure depression, which is associated with smell dysfunction. Participants will answer questions about how they are feeling and how ready they are to contact a healthcare provider. The specific smell tests that will be given to participants will be either SCENTinel, NIH Toolbox, Arohma, or the B-SIT test. Other Follow-Up Questions include ones regarding access to care, contacting a provider, seeing a provider, and satisfaction with care.

ELIGIBILITY:
Inclusion Criteria:

- Can read and understand English and have access to a reliable internet connection and a smart device or computer for the duration of the experimental sessions, unless they are part of community events in which smart devices are provided

Exclusion Criteria:

- Known intolerance or allergy to any of the odor stimuli used

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Measuring depression symptoms using the PHQ-9 score | PHQ-9 is completed at baseline, during 1 month follow-up session, and during the 6 month follow-up.
  The PHQ-9 is a screening measure of depressive symptoms.

SECONDARY OUTCOMES:
Measuring health-related quality of life using the SF-12 survey. | SF-12 is completed at baseline, during 1 month follow-up session, and during the 6 month follow-up.
  The SF-12 is a screening measure of health-related quality of life.
Measuring self-reported health perception using a "How do you feel?" 0-100 Visual Analogue Scale (VAS). | VAS is completed at baseline, during 1 month follow-up session, and during the 6 month follow-up.
  "How do you feel?" VAS is a self-reported measure of health perception.
Effectiveness of implementation (to contact a healthcare provider for smell dysfunction within up to 6 months from smell testing). | Evaluated during 1 month and 6 month follow ups
  Participants are asked a Yes or No question about whether they contacted a healthcare provider. The investigators will examine the proportion of participants connecting with a healthcare provider for smell dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Parma, Principal Investigator — Monell Chemical Senses Center; Pamela Dalton, Principal Investigator — Monell Chemical Senses Center; Danielle Reed, Principal Investigator — Monell Chemical Senses Center
Locations (1):
- Monell Chemical Senses Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected data
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: When data collection begins, it will be uploaded to Hub4Smell and available for accessing following completion of data collection for every 250 participants. Once access to data on Hub4Smell has been granted, data will be available indefinitely.
Access Criteria: Study subject data will be anonymized before data upload to the Hub4Smell database. The anonymization algorithm will be shared with the Hub4Smell Contributors by the Hub4Smell leadership team. Internally, Hub4Smell will associate a persistent surrogate key to identify each record. The study will include metadata attributes to define the data that will be shared with the Hub4Smell database. The Hub4Smell leadership team will trigger loading and sharing procedures of data to the Hub4Smell database. Data will be loaded privately and when marked ready to be shared, will become available to the Hub4Smell Contributors, who will be informed that a new batch of data has been uploaded. Consumers of the data will be required to create an account to download data. Access to source code will be controlled through GitHub user accounts. Access will be approved by the multiple principal investigators (MPIs) and technical teams. Data will be available indefinitely at this time.